CLINICAL TRIAL: NCT04977050
Title: Keeping Rural Minority 'Essential' Workplaces Open Safely During the COVID-19 Pandemic: The Role of Frequent Point-of-care Molecular Workplace Surveillance for Miners (Short Title: The Miners' Pandemic Project)
Brief Title: The Role of Frequent Point-of-care Molecular Workplace Surveillance for Miners
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HRPO 20-680; 3U01GM132175-03S1 (NIH)
Record Dates: First submitted 2021-07-14; First posted 2021-07-26 (Actual); Results first posted 2024-04-03 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Two groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Site (Experimental): All miners in the New Mexico intervention mine site who will be administered nasal swabs for antigen testing every other work shift, and serological testing 3 months.
  Interventions: Diagnostic Test: Quidel quickvue antigen test for COVID-19
- Controled site (No Intervention): All miners in the Wyoming Control mine site who will be administered serological testing 3 months.

INTERVENTIONS:
Diagnostic Test: Quidel quickvue antigen test for COVID-19 — rapid antigen test on nasal swab specimen for COVID-19
  Arms: Intervention Site

SUMMARY:
The long-term goal of the study is to mitigate the spread of the pandemic in miners, a population of high-risk, rural essential workers who are susceptible and vulnerable to COVID-19, partly based on exposure to particulate air pollution, and who are predominantly racial/ethnic minorities in New Mexico (NM) (3, 11). The study objective is to provide proof-of-principle for frequent point-of-care molecular testing as a workplace surveillance tool to monitor and prevent the spread of SARS-CoV-2 infection in this unique population. The central hypothesis is that frequent workplace molecular surveillance is an effective method to reduce SARS-CoV-2 infection and discover novel host risk factors for the virus. The site of molecular surveillance (intervention site) will be a surface coal mine in McKinley County, NM, located just outside the Eastern Agency of the Navajo Nation, comprised of 66% minority miners. This site offers a unique opportunity for a community-based study of SARS-CoV-2 infection in this population. Miners at the intervention site will provide nasal swabs before beginning their work shift on alternate days that will be analyzed with a 'screening' molecular test (12). This test is ideal because it is low cost, simple, portable, point-of-care, rapid, and can be performed by minimally trained professionals in low-infrastructure settings. The control site is a similar coal mine in Campbell County, Wyoming (WY). Both mines, operated by the same company, have similar engineering, administrative, and personal protective measures in place. The rationale for this study is to establish the suitability of longitudinal molecular surveillance to prevent and control SARS-CoV-2 infection in this unique population by completing the following specific aims.

DETAILED DESCRIPTION:
Specific Aim 1: To determine the acceptance rate to frequent point-of-care molecular workplace surveillance among miners.

Hypothesis 1: Miners will have a cumulative acceptance rate of frequent testing at ≥85%, with the added objective of exploring difference in acceptance by miner characteristics.

Specific Aim 2: To determine the ability to detect the presence of SARS-CoV-2 by point-of-care molecular workplace surveillance in a real-world setting of miners.

Hypothesis 2: The sensitivity of the screening test in a real-world study setting is a) comparable to that described by others in controlled settings, and b) positively associated with viral load in upper respiratory specimens (latter measured in nose and nasopharynx using quantitative reverse transcriptase-polymerase chain reaction or RT-PCR).

Specific Aim 3: To determine the effectiveness and implementation costs of frequent point-of-care molecular workplace surveillance on reducing incident infection rates of SARS-CoV-2.

Hypothesis 3A: Frequent point-of-care molecular testing over six months in the intervention mine will result in lower incident seropositivity rates compared to the control mine.

Hypothesis 3B: Frequent point-of-care molecular surveillance in the intervention mine is cost-effective compared to the control mine.

Specific Aim 4: To determine novel predictive host factors associated with incident SARS-CoV-2 infection in miners.

Hypothesis 4: Miners with incident infection demonstrate less frequent use of cloth face-coverings outside the workplace, greater mine dust exposure intensity, presence of dust-related lung disease, and racial/ethnic minority status than those not infected.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female Miner employed at intervention mine or the control mine.
* > 18 years of age.
* Willing and able to provide and sign Informed Consent Form.
* Willing and able to comply with study procedures.

Exclusion Criteria:

* Unable or unwilling to provide and sign Informed Consent Form
* < 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aksay Sood, MD, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: Yes
Plan to share with Duke Clinical Research Institute. As per NIH requirements.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: from current to Infinite
Access Criteria: request to Duke Clinical Research Institute

REFERENCES:
- [Background] Sood A, Pollard C, Suer KL, Vlahovich K, Walker J. Caring for Miners During the Coronavirus Disease-2019 (COVID-19) Pandemic. J Rural Health. 2021 Jan;37(1):165-168. doi: 10.1111/jrh.12444. Epub 2020 Jun 2. No abstract available. PMID 32277775
- [Derived] Constantin AM, Noertjojo K, Sommer I, Pizarro AB, Persad E, Durao S, Nussbaumer-Streit B, McElvenny DM, Rhodes S, Martin C, Sampson O, Jorgensen KJ, Bruschettini M. Workplace interventions to reduce the risk of SARS-CoV-2 infection outside of healthcare settings. Cochrane Database Syst Rev. 2024 Apr 10;4(4):CD015112. doi: 10.1002/14651858.CD015112.pub3. PMID 38597249

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention Site | Controled Site
Started | 169 | 61
Completed | 169 | 61
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Site | Controled Site | Total
Number analyzed (Participants) | 169 | 61 | 230
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 13 | 0 | 13
  Between 18 and 65 years | 154 | 60 | 214
  >=65 years | 2 | 1 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (11.2) | 45.2 (11.9) | 44.6 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 3 participants opted to not report or reported as intersex.
  Participants
    number analyzed (Participants) | 168 | 59 | 227
    Female | 14 | 11 | 25
    Male | 154 | 48 | 202
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 97 | 4 | 101
  Not Hispanic or Latino | 63 | 54 | 117
  Unknown or Not Reported | 9 | 3 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 27 | 2 | 29
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 96 | 56 | 152
  More than one race | 31 | 3 | 34
  Unknown or Not Reported | 14 | 0 | 14
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 169 | 61 | 230

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Screened (Molecular)
Description: Rapid antigen test for COVID-19
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Site | Controled Site
Number analyzed (Participants) | 169 | 61
Participants | 169 | 61

ADVERSE EVENTS:
Time Frame: 1 year
Description: Study was data collection. Nasal swab and serology testing is low risk.
Arm/Group | Intervention Site | Controled Site
All-Cause Mortality (participants affected / at risk) | 0/169 | 0/61
Serious Adverse Events (participants affected / at risk) | 0/169 | 0/61
Other Adverse Events (participants affected / at risk) | 0/169 | 0/61

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-15): https://cdn.clinicaltrials.gov/large-docs/50/NCT04977050/Prot_SAP_000.pdf